CLINICAL TRIAL: NCT01546779
Title: The Immediate Effect of Resistive Expiration Via "Volumetric Incentive Spirometer" on Lung Function in Patients With Cystic Fibrosis.
Brief Title: The Use of Visual Feedback in Airway Clearance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-08-5583-OE-CTIL
Record Dates: First submitted 2012-02-19; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lung function (Experimental)
  Interventions: Device: Tri-Gym

INTERVENTIONS:
Device: Tri-Gym — 40 CF patients performed airway clearance using the VISex, by exhaling against chosen resistance being motivated by visual feedback of raising colored balls. The level of resistance was set to cause longest expiration/volume, until mucus was transported from the peripheral to the central airways, to be expectorated by the subsequent cough.
  Other Names: incentive spirometer

SUMMARY:
Cystic Fibrosis (CF) patients perform airway clearance incorporating various breathing strategies, to clear secretions from their lungs. Hand held devices may aid mucus expectoration, and also motivate the patient to manage by themselves. Our aims was to study if resistive expiration through "volumetric incentive spirometer" (VISex) can improve lung function in the short term in Cystic Fibrosis (CF) patients.

ELIGIBILITY:
Inclusion Criteria:

* cystic fibrosis patients

Exclusion Criteria:

* i.v. antibiotic therapy during the experiment day

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
lung function | fifteen minutes after intervention
  Forced expiratory maneuvers were measured before and 15 minutes after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- The Pediatric Pulmonary Unit the Edmond and LiliSafraChildrens Hospital, Sheba Medical Center, Ramat Gan, Israel, Israel